CLINICAL TRIAL: NCT06174142
Title: A Randomized Controlled Trial Comparing Two Protocols of Shock Wave Therapy for Patients With Plantar Fasciitis
Brief Title: Comparing Two Protocols of Shock Wave Therapy for Patients With Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Fatima Alkalbani, Student, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAlkalbani
Record Dates: First submitted 2023-11-09; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: This randomized trial compares two shock wave therapy protocols in plantar fasciitis treatment against a sham control. Group A receives high-frequency therapy (15 Hz, intensity level 3), Group B low-frequency (10 Hz, intensity level 4), and Group C a sham treatment, all alongside physical therapy. The goal is to evaluate pain reduction and functional improvement after six sessions, with follow-up assessments to gauge effect durability.
Who Masked: Participant
Masking Description: In a randomized trial, two shock wave therapies for plantar fasciitis are tested. Group A gets high-frequency (15 Hz), Group B low-frequency (10 Hz, higher intensity), and Group C receives sham therapy. The study aims to measure pain relief and functional gains post six treatments, with follow-ups to assess benefits' persistence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Frequency ESWT Group (Experimental): This arm will receive extracorporeal shockwave therapy (ESWT) with a higher frequency setting of 15 Hz and an intensity/pressure of level 3. Participants will receive a total of 1800 impulses per session for 6 sessions, with one session per week, alongside a selected physical therapy program.
  Interventions: Device: High-Frequency ESWT
- Low-Frequency ESWT Group (Experimental): Experimental
  Interventions: Device: Low-Frequency ESWT Group
- Sham ESWT Control Group (Sham Comparator): Participants in the control group will undergo a sham shockwave therapy protocol, which simulates ESWT treatment without actual therapeutic effects, to serve as a comparison for the active treatments. They will also engage in the same physical therapy program as the other two arms.
  Interventions: Device: Sham ESWT Control Group

INTERVENTIONS:
Device: High-Frequency ESWT — Participants will receive extracorporeal shock wave therapy at a frequency of 15 Hz and intensity/pressure level 3, with a total of 1800 impulses per session. This intervention will be conducted once per week for six weeks, alongside a standard physical therapy regimen
  Arms: High-Frequency ESWT Group
Device: Low-Frequency ESWT Group — "Participants will be treated with extracorporeal shock wave therapy at a frequency of 10 Hz and intensity/pressure level 4, also with a total of 1800 impulses per session. This protocol will be delivered weekly for six sessions, accompanied by standardized physical therapy exercises."
  Arms: Low-Frequency ESWT Group
Device: Sham ESWT Control Group — "Participants in this control group will undergo a sham ESWT procedure that mimics the treatment experience without actual therapeutic effects, ensuring the blinding of participants. This sham therapy will be scheduled once a week for six weeks, in conjunction with the same physical therapy program as the other groups."
  Arms: Sham ESWT Control Group

SUMMARY:
The goal of this clinical trial is to compare the efficacy of two distinct shock wave therapy protocols and their impact on improving function and reducing pain in individuals with plantar fasciitis, a common cause of heel pain that affects millions worldwide.

The key questions the study aims to address are:

How effective is each shock wave therapy protocol in enhancing functional ability without pain in patients with plantar fasciitis? Does either protocol offer a significant benefit over the other in terms of pain relief and functional improvement after a course of six treatment sessions?

Participants will be randomly assigned to one of three groups and will engage in the study as follows:

Undergo six sessions of shock wave therapy with parameters specific to their assigned group.

Complete questionnaires assessing foot function and pain levels. Participate in evaluations before, during, and after the treatment to monitor their progress.

The three groups in the comparison are as follows:

Group A will receive shock wave therapy at a higher frequency and specific intensity, with a set number of impulses.

Group B will undergo therapy with a different frequency and intensity level but will receive the same number of impulses.

Group C, the control group, will receive a sham therapy, mirroring the treatment experience without the therapeutic effects to serve as a baseline for comparison.

The study is anticipated to delineate a more effective protocol for treating plantar fasciitis with shock wave therapy. The findings may contribute to enhanced treatment guidelines, potentially resulting in faster recovery times for patients. The participation of individuals in this research will offer valuable insights that could inform future therapeutic strategies for managing plantar fasciitis

DETAILED DESCRIPTION:
This randomized controlled trial is designed to evaluate the efficacy of two distinct shock wave therapy protocols in treating plantar fasciitis, a condition that causes heel pain and can severely impact daily activities. The aim is to discern which protocol is more effective at improving functional abilities and reducing pain.

Plantar fasciitis typically manifests as a sharp pain at the bottom of the heel, often affecting individuals who engage in high-impact activities such as running. With the variability in treatment approaches, shock wave therapy has been recognized as a promising, non-invasive treatment method. The study seeks to address the current gaps in research by identifying the most beneficial treatment parameters of shock wave therapy.

Participants will be randomly allocated to one of three groups:

Group A will receive shock wave therapy with high-frequency settings. Group B will receive shock wave therapy with low-frequency settings but higher intensity.

Group C will serve as a control group, receiving sham shock wave therapy to provide a baseline for comparison.

All groups will partake in a consistent regimen of physical therapy exercises, ensuring that any differences in outcomes are attributable to the shock wave therapy parameters. The inclusion of these exercises is crucial as they contribute to recovery by stretching and strengthening the affected area.

To maintain the integrity of the trial, participants will be blinded to the shock wave therapy parameters they receive, thereby reducing potential bias. The study will feature comprehensive assessments at various points: before the intervention, halfway through the sessions, upon completion of the therapy, and during a follow-up phase to assess the durability of the effects.

The trial is anticipated to yield significant insights into the effectiveness of different shock wave therapy protocols, which will be instrumental in developing more refined treatment guidelines. Ultimately, these findings could enhance the quality of life for individuals with plantar fasciitis and guide clinical practice for the treatment of associated heel pain.

ELIGIBILITY:
Inclusion Criteria:

1. The participants should present with unilateral pain
2. The participants' age will be ranged from 20-50 years old.
3. The participants should have the pain from for at least 6 weeks.
4. Moderate disability as assessed by the foot function index (FFI)
5. The Body Mass Index (BMI) should be normal.
6. The participants should have pronated feet (6-9 on the foot posture index)

Exclusion Criteria:

1. History of surgery or fracture
2. History of corticosteroid injection within 6 months
3. Unable to follow or understand the instructions
4. High BMI
5. Severe foot pronation (+10 on the foot posture index)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-01-05 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | Baseline: Assessment before the start of intervention (Week 0). Mid-Point: After the 3rd session (end of Week 3). End of Treatment: After the 6th session (end of Week 6). Follow-Up: 12 weeks post-intervention (end of Week 18).
  Evaluate the decrease in heel pain as measured by the Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Functional Improvement | Baseline: Assessment before the start of intervention (Week 0). Mid-Point: After the 3rd session (end of Week 3). End of Treatment: After the 6th session (end of Week 6). Follow-Up: 12 weeks post-intervention (end of Week 18).
  Measure the change in foot function using the Foot Function Index (FFI).

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Alkalbani, Bsc, Principal Investigator — PRS User

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data collected during this trial outside of the study team and the immediate research purposes outlined in the protocol. Data sharing decisions will be revisited upon study completion and publication of results, considering participant consent, data sensitivity, and ethical considerations

REFERENCES:
- [Background] Riddle DL, Schappert SM. Volume of ambulatory care visits and patterns of care for patients diagnosed with plantar fasciitis: a national study of medical doctors. Foot Ankle Int. 2004 May;25(5):303-10. doi: 10.1177/107110070402500505. PMID 15134610
- [Background] Dunn JE, Link CL, Felson DT, Crincoli MG, Keysor JJ, McKinlay JB. Prevalence of foot and ankle conditions in a multiethnic community sample of older adults. Am J Epidemiol. 2004 Mar 1;159(5):491-8. doi: 10.1093/aje/kwh071. PMID 14977645
- [Background] Petraglia F, Ramazzina I, Costantino C. Plantar fasciitis in athletes: diagnostic and treatment strategies. A systematic review. Muscles Ligaments Tendons J. 2017 May 10;7(1):107-118. doi: 10.11138/mltj/2017.7.1.107. eCollection 2017 Jan-Mar. PMID 28717618
- [Background] Leao RG, Azuma MM, Ambrosio GHC, Faloppa F, Takimoto ES, Tamaoki MJS. Effectiveness of shockwave therapy in the treatment of plantar fasciitis. Acta Ortop Bras. 2020 Jan-Feb;28(1):7-11. doi: 10.1590/1413-785220202801227402. PMID 32095104
- [Background] Xu D, Jiang W, Huang D, Hu X, Wang Y, Li H, Zhou S, Gan K, Ma W. Comparison Between Extracorporeal Shock Wave Therapy and Local Corticosteroid Injection for Plantar Fasciitis. Foot Ankle Int. 2020 Feb;41(2):200-205. doi: 10.1177/1071100719891111. Epub 2019 Nov 19. PMID 31744313
- [Background] Luffy L, Grosel J, Thomas R, So E. Plantar fasciitis: A review of treatments. JAAPA. 2018 Jan;31(1):20-24. doi: 10.1097/01.JAA.0000527695.76041.99. PMID 29227320
- [Background] Schwartz EN, Su J. Plantar fasciitis: a concise review. Perm J. 2014 Winter;18(1):e105-7. doi: 10.7812/TPP/13-113. PMID 24626080
- [Background] Thompson JV, Saini SS, Reb CW, Daniel JN. Diagnosis and management of plantar fasciitis. J Am Osteopath Assoc. 2014 Dec;114(12):900-6. doi: 10.7556/jaoa.2014.177. PMID 25429080
- [Background] Lemont H, Ammirati KM, Usen N. Plantar fasciitis: a degenerative process (fasciosis) without inflammation. J Am Podiatr Med Assoc. 2003 May-Jun;93(3):234-7. doi: 10.7547/87507315-93-3-234. PMID 12756315
- [Background] Gollwitzer H, Saxena A, DiDomenico LA, Galli L, Bouche RT, Caminear DS, Fullem B, Vester JC, Horn C, Banke IJ, Burgkart R, Gerdesmeyer L. Clinically relevant effectiveness of focused extracorporeal shock wave therapy in the treatment of chronic plantar fasciitis: a randomized, controlled multicenter study. J Bone Joint Surg Am. 2015 May 6;97(9):701-8. doi: 10.2106/JBJS.M.01331. PMID 25948515
- [Background] Rompe JD, Decking J, Schoellner C, Nafe B. Shock wave application for chronic plantar fasciitis in running athletes. A prospective, randomized, placebo-controlled trial. Am J Sports Med. 2003 Mar-Apr;31(2):268-75. doi: 10.1177/03635465030310021901. PMID 12642264
- [Background] Garrett TR, Neibert PJ. The effectiveness of a gastrocnemius-soleus stretching program as a therapeutic treatment of plantar fasciitis. J Sport Rehabil. 2013 Nov;22(4):308-12. doi: 10.1123/jsr.22.4.308. Epub 2013 May 22. PMID 23752554
- [Background] Thong-On S, Bovonsunthonchai S, Vachalathiti R, Intiravoranont W, Suwannarat S, Smith R. Effects of Strengthening and Stretching Exercises on the Temporospatial Gait Parameters in Patients With Plantar Fasciitis: A Randomized Controlled Trial. Ann Rehabil Med. 2019 Dec;43(6):662-676. doi: 10.5535/arm.2019.43.6.662. Epub 2019 Dec 31. PMID 31918529
- [Background] Cheing GL, Chang H. Extracorporeal shock wave therapy. J Orthop Sports Phys Ther. 2003 Jun;33(6):337-43. doi: 10.2519/jospt.2003.33.6.337. No abstract available. PMID 12839209
- [Background] Budiman-Mak E, Conrad KJ, Roach KE. The Foot Function Index: a measure of foot pain and disability. J Clin Epidemiol. 1991;44(6):561-70. doi: 10.1016/0895-4356(91)90220-4. PMID 2037861
- [Background] Saag KG, Saltzman CL, Brown CK, Budiman-Mak E. The Foot Function Index for measuring rheumatoid arthritis pain: evaluating side-to-side reliability. Foot Ankle Int. 1996 Aug;17(8):506-10. doi: 10.1177/107110079601700814. PMID 8863033
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293